CLINICAL TRIAL: NCT06948552
Title: A Phase II Study on Photodynamic Diagnosis of Urological Cancer in the Upper Urinary Tract Using Fluorescence Endoscopy With Cystoscopy and Ureteroscopy With 5-ALA
Brief Title: Photodynamic Diagnosis of Upper Tract Urothelial Carcinoma Using Fluorescence Endoscopy and Oral 5-ALA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Johar Raza, Urologic Oncologist, Henry Ford Health, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HFH-IRB17325; IRB17325 (Other: Henry Ford Health IRB)
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Upper Tract Urothelial Carcinoma
Keywords: Photodynamic Diagnosis; 5-ALA; Gleolan; Ureteroscopy; Fluorescence Endoscopy; Urothelial Cancer; Blue Light; Kidney Cancer; Urologic Oncology; Minimally Invasive Surgery
MeSH Terms: conditions — Kidney Neoplasms | interventions — Aminolevulinic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- 5-ALA Fluorescence Imaging (Experimental): Participants will receive a single oral dose of 5-aminolevulinic acid (5-ALA, Gleolan) 2-4 hours prior to ureteroscopic tumor resection. Blue light endoscopy will be used intraoperatively to assess tumor fluorescence and aid in visualization and resection.
  Interventions: Drug: 5-Aminolevulinic acid Hydrochloride (Gliolan®)

INTERVENTIONS:
Drug: 5-Aminolevulinic acid Hydrochloride (Gliolan®) — Participants will receive a single oral dose of 5-aminolevulinic acid (20 mg/kg) approximately 2 to 4 hours prior to surgery. The goal is to evaluate the feasibility of using fluorescence cystoscopy with blue light to improve tumor detection and visualization during ureteroscopic resection of upper tract urothelial carcinoma.

SUMMARY:
This study is evaluating whether a medication called 5-aminolevulinic acid (5-ALA), approved by the FDA for use in brain surgery, can help improve the visibility of upper tract urothelial tumors during surgery. Patients undergoing ureteroscopic tumor resection will receive 5-ALA prior to surgery, and surgeons will use special blue light to help identify abnormal tissue that might not be seen under standard white light. The goal is to assess whether this technique can enhance tumor detection and removal.

DETAILED DESCRIPTION:
This is a prospective, single-arm feasibility study investigating the use of 5-aminolevulinic acid (5-ALA, Gleolan) to enhance intraoperative tumor visualization in patients undergoing ureteroscopic resection for suspected upper tract urothelial carcinoma (UTUC). 5-ALA is an FDA-approved oral agent used in glioma surgery to promote fluorescence of malignant tissue under blue light. This study will evaluate whether similar visualization can be achieved in the upper urinary tract to aid in the identification and resection of UTUC. Up to 10 participants will be enrolled. Safety, technical feasibility, and tumor detection outcomes will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or older undergoing diagnostic or therapeutic ureteroscopy for a known or suspected upper tract urothelial tumor
* Able to provide informed consent
* Able to comply with study requirements

Exclusion Criteria:

* Known porphyria or hypersensitivity to porphyrins
* Pregnant or breastfeeding women
* AST or ALT > 2x upper limit of normal within 30 days prior to surgery
* Participation in another investigational study within 30 days
* Known allergy or contraindication to 5-ALA or its components

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Detection of tumor fluorescence using 5-ALA under blue light | Day of Surgery
  Surgeons will assess whether upper tract urothelial tumors exhibit visible fluorescence under blue light following oral administration of 5-ALA (20 mg/kg). Presence or absence of fluorescence will be recorded for each lesion during ureteroscopic resection.

SECONDARY OUTCOMES:
Incidence and severity of adverse events following 5-ALA administration | Up to 30 days post-procedure
  Participants will be monitored for any adverse events following oral 5-ALA administration. Events will be assessed using CTCAE v5.0 criteria, with specific focus on known side effects such as nausea, vomiting, hypotension, and photosensitivity reactions. Lab abnormalities and any serious adverse events will also be documented.
Presence of residual tumor at follow-up ureteroscopy | Up to 3 months post-procedure
  For patients who undergo a second-look ureteroscopy within 3 months of initial resection, surgeons will assess for visible tumor at the prior resection sites. Findings will be used to evaluate the completeness of initial resection and the potential benefit of 5-ALA fluorescence guidance.

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
This is a single-site, investigator-initiated feasibility study funded through an internal philanthropic research grant. Individual participant data will not be shared, as there is no formal data-sharing infrastructure in place and the study is not intended to support regulatory submissions or external data analysis.

REFERENCES:
- [Background] Taoka R, Matsuoka Y, Yamasaki M, Kani N, Honda T, Harada S, Tohi Y, Kato T, Okazoe H, Tsunemori H, Ueda N, Sugimoto M. Photodynamic diagnosis-assisted transurethral resection using oral 5-aminolevulinic acid decreases residual cancer and improves recurrence-free survival in patients with non-muscle-invasive bladder cancer. Photodiagnosis Photodyn Ther. 2022 Jun;38:102838. doi: 10.1016/j.pdpdt.2022.102838. Epub 2022 Apr 4. PMID 35381368
- [Background] Watanabe K, Tamura K, Matsushita Y, Watanabe H, Motoyama D, Ito T, Sugiyama T, Otsuka A, Miyake H. Significance of 5-Aminolevulinic Acid-mediated Photodynamic Diagnosis Following Standard Transurethral Resection in Non-muscle Invasive Bladder Cancer. Cancer Diagn Progn. 2021 Jul 3;1(3):201-205. doi: 10.21873/cdp.10027. eCollection 2021 Jul-Aug. PMID 35399308
- [Background] Nakai Y, Inoue K, Tsuzuki T, Shimamoto T, Shuin T, Nagao K, Matsuyama H, Oyama M, Furuse H, Ozono S, Miyake M, Fujimoto K. Oral 5-aminolevulinic acid-mediated photodynamic diagnosis using fluorescence cystoscopy for non-muscle-invasive bladder cancer: A multicenter phase III study. Int J Urol. 2018 Aug;25(8):723-729. doi: 10.1111/iju.13718. Epub 2018 Jul 12. PMID 29999205
- [Background] Yoshida T, Setsuda S, Ishizuka M, Inoue T, Kinoshita H, Matsuda T. Photodynamic Diagnosis with Oral 5-Aminolevulinic Acid for Upper Urinary Tract Carcinoma: A Prospective Clinical Trial. J Endourol. 2020 Apr;34(4):509-515. doi: 10.1089/end.2019.0725. Epub 2020 Mar 31. PMID 31964177
- [Background] Fukuhara H, Kurabayashi A, Furihata M, Setuda S, Takahashi K, Murakami K, Tanaka T, Inoue K. 5-aminolevulinic acid-mediated photodynamic diagnosis using fluorescence ureterorenoscopy for urinary upper tract urothelial carcinoma approximately Preliminary prospective single centre trial approximately . Photodiagnosis Photodyn Ther. 2020 Mar;29:101617. doi: 10.1016/j.pdpdt.2019.101617. Epub 2019 Dec 16. PMID 31857216
- See also: Primary FDA Approval Citation — https://www.fda.gov/drugs/resources-information-approved-drugs/aminolevulinic-acid-hydrochloride-known-ala-hcl-gleolan-nx-development-corp-optical-imaging-agent